CLINICAL TRIAL: NCT06192940
Title: Impact of Smart Connected Insulin Pens on Quality of Life in Dependent Patients with Diabetes Using Continuous Glucose Measurement
Acronym: BESTYLCO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0052
Record Dates: First submitted 2023-12-07; First posted 2024-01-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
Keywords: insulin practice; Dependent patient; Smart connected insulin pen
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Counseling home caregivers — Advice on the proper use of insulin therapy will be given, if necessary, to caregivers. Patients are reviewed at 1 month of this first visit with a collection of the same data

SUMMARY:
Insulin-treated diabetes in dependent or institutionalized patients is often poorly balanced and continuous glucose measurement is underused. The purpose of this tudy is to know how smart connected insulin pens and continuous glucose measurement can improve insulin therapy practice in dependent and/or institutionalized patients?

DETAILED DESCRIPTION:
Insulin-treated diabetes in dependent or institutionalized patients is often poorly balanced and continuous glucose measurement is underused. Current practice and my experience in diabetes show a misuse of insulin therapy by caregivers at home and in institutions. Studies on the elderly insulin-treated person living in institutions show, through continuous glucose measurement, frequent nocturnal hypoglycemia at 79%. The continuous measurement of glucose has also shown its interest in reducing hospitalizations for acute event and, permanently.

A norwegian study shows that hypoglycemic treatments are too frequently prescribed in nursing homes. Hospitalizations for severe hypoglycemia are often due to dose errors or unsupervised recommendations in people over 65 years.

Smart connected insulin pens have shown a benefit in the management of insulin therapy in patients living with type 1 diabetes, improving glycemic balance.

Study focuses on the identification of misuses of insulin therapy in dependent and/or institutionalized patients. A study of everyday life, we expect a decrease in dysfunctions in patients equipped with a continuous glucose measurement system and connected pens after advice given to their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years patient with type 1 or 2 diabetes
* Treated with multiple insulin injections
* Equipped with a continuous glucose measurement system and smart connected insulin pens at least one month before
* Dependent on a health professional for treatment management.
* Subject informed of the study and not objecting to data collection.

Exclusion Criteria:

- Patient refusing study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient managed by a caregivers for the management of insulin therapy at home or in nursing home or in healthcare facility.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin Injection | at day 0
  Percentage of insulin injections not as prescribed

SECONDARY OUTCOMES:
number of missed injections | at day 0
  Percentage of missed injections
number of injections | at day 0
  Percentage of injections performed with a dose deviation of +-20% from the prescribed dose
number of injections | at day 0
  Percentage of injections performed outside the meal time : more than 15 minutes before or more than an hour after the meal.
Continuous glucose measurement parameters | at day 0
  Time in range
Continuous glucose measurement parameters | at day 30
  Time in range
Acute Diabetes Events | at day 0
  severe hypoglycemia, hyperglycemia requiring hospitalization
Acute Diabetes Events | at day 30
  severe hypoglycemia, hyperglycemia requiring hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Marie BOULY, APN, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouillet B, Tscherter P, Vaillard L, Nonciaux C, Hourdain P, Ravier A, Rouland A, Petit JM, Verges B, Quilot E. Frequent and severe hypoglycaemia detected with continuous glucose monitoring in older institutionalised patients with diabetes. Age Ageing. 2021 Nov 10;50(6):2088-2093. doi: 10.1093/ageing/afab128. PMID 34324624
- [Background] Guerci B, Roussel R, Levrat-Guillen F, Detournay B, Vicaut E, De Pouvourville G, Emery C, Riveline JP. Important Decrease in Hospitalizations for Acute Diabetes Events Following FreeStyle Libre System Initiation in People with Type 2 Diabetes on Basal Insulin Therapy in France. Diabetes Technol Ther. 2023 Jan;25(1):20-30. doi: 10.1089/dia.2022.0271. Epub 2022 Nov 24. PMID 36094418
- [Background] Riveline JP, Roussel R, Vicaut E, de Pouvourville G, Detournay B, Emery C, Levrat-Guillen F, Guerci B. Reduced Rate of Acute Diabetes Events with Flash Glucose Monitoring Is Sustained for 2 Years After Initiation: Extended Outcomes from the RELIEF Study. Diabetes Technol Ther. 2022 Sep;24(9):611-618. doi: 10.1089/dia.2022.0085. Epub 2022 Jul 11. PMID 35604792
- [Background] Andreassen LM, Sandberg S, Kristensen GB, Solvik UO, Kjome RL. Nursing home patients with diabetes: prevalence, drug treatment and glycemic control. Diabetes Res Clin Pract. 2014 Jul;105(1):102-9. doi: 10.1016/j.diabres.2014.04.012. Epub 2014 Apr 28. PMID 24853809
- [Background] Poret F, Nacher M, Pujo J, Cauvin JM, Demar M, Massicard M, Sabbah N. Risk factors for hypoglycaemia in people with diabetes admitted to the Emergency Department of a Hospital in French Guiana. Diabet Med. 2022 Feb;39(2):e14736. doi: 10.1111/dme.14736. Epub 2021 Nov 23. PMID 34738244
- [Background] Ekberg NR, Hartvig NV, Kaas A, Moller JB, Adolfsson P. Smart Pen Exposes Missed Basal Insulin Injections and Reveals the Impact on Glycemic Control in Adults With Type 1 Diabetes. J Diabetes Sci Technol. 2024 Jan;18(1):66-73. doi: 10.1177/19322968221104142. Epub 2022 Jul 1. PMID 35775735
- [Background] Coleman BJ. European models of long-term care in the home and community. Int J Health Serv. 1995;25(3):455-74. doi: 10.2190/FYP6-DLWY-WKKT-6NNJ. PMID 7591375